CLINICAL TRIAL: NCT03942081
Title: Testing the Accuracy and Feasibility of Diabetic Foot Ulcer Imaging
Brief Title: Diabetic Foot Ulcer Imaging- Study 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linnea Polgreen (Other)
Collaborators: Fraternal Order of the Eagles Diabetes Research Center (Unknown)
Responsible Party: Sponsor-Investigator, Linnea Polgreen, Associate Professor, Department of Pharmacy Practice and Science / Division of Health Services Research, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 201706725
Record Dates: First submitted 2019-05-06; First posted 2019-05-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Foot Ulcer; Foot Ulcer, Diabetic
MeSH Terms: conditions — Foot Ulcer; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Ulcer Measurement and Photo Group (Experimental): Diabetic patients with foot ulcers being seen in clinic.
  Interventions: Device: Ulcer Measurement Software
- Healthy Control Group (No Intervention): Patients without foot ulcers being seen in the clinic.

INTERVENTIONS:
Device: Ulcer Measurement Software — Photos being taken of foot ulcers. Software estimation of foot ulcer being compared to actual measured size.
  Arms: Ulcer Measurement and Photo Group

SUMMARY:
All study procedures will occur during one appointment. The research team will measure the size of the foot ulcer (if one is present) and multiple photos will be taken with a smart phone camera and thermal camera. Demographic information will be obtained from the medical record.

DETAILED DESCRIPTION:
The research procedures consist of a) a research assistant measuring the size of the foot ulcer (for ulcer patients), b) patients having pictures of their feet taken with a smart phone under 4 conditions- 1) photos taken by researchers, 2) photos taken by the patient by hand, 3) photos taken by the patient with a selfie stick, and 4) photos taken by a 3rd party (e.g., friend/family member of patient). If the patient is not able to take photographs under any of the conditions, that condition will be excluded. In addition to photos being taken with a smart phone, additional photos will be taken with a thermal camera by the research team to determine if there is a difference in ulcer size depending on type of camera used. It is anticipated that procedures will last between 15 and 45 minutes. There is no long-term follow-up. If a patient returns to the clinic they will be asked if they wish to complete all study procedures again. Once the patient has left the clinic, the research team will check the medical record for: age, sex, race, ethnicity, BMI, co-morbidities, and zip code (to determine if patient lives in an urban or rural location).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 1 or Type 2 Diabetes
* Has a current foot lesion
* Receiving care through University of Iowa Hospitals and Clinics (UIHC) Iowa River Landing Diabetes Clinic, UIHC Internal Medicine Clinic, or UIHC Orthopedic Clinic.

Exclusion Criteria:

* Cognitive impairment that prevents consent
* Lack of fluency in speaking or understanding English
* Known aversion to research studies

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Foot Ulcer Size | 45 minutes
  Size of foot ulcers will be determined by measurement and estimated by software

SECONDARY OUTCOMES:
Quality of Photos: 1 - 5 scale | 45 minutes
  Quality of foot ulcer photos will be quantitatively assessed using a 1 - 5 scale (with 1 being poor focus and lighting and 5 being excellent focus and lighting). These scores will be determined subjectively by multiple researchers and averaged to a single score.

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Polgreen, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No